CLINICAL TRIAL: NCT06283225
Title: Pilot Study to Investigate the Influence of a Dysmenorrhoea App on the Quality of Life and Symptoms of Patients
Brief Title: Pilot Study to Investigate the Effect of a Dysmenorrhoea App
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endo Health GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RCT004_PilotPia
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Dysmenorrhea
Keywords: digital; app; dysmenorrhea; quality of life
MeSH Terms: conditions — Dysmenorrhea; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: intervention group and control group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): the intervention group has access to the dysmenorrhoea app and its functions in addition to normal regular care.
  Interventions: Device: Pia-App
- Control group (No Intervention): the intervention group has access to normal regular care only.

INTERVENTIONS:
Device: Pia-App — The dysmenorrhoea app (Pia-App) is evidence-based and helps patients to implement continuous multimodal (pain) treatment that is integrated into everyday life. Symptoms, events, influencing factors and examinations can be recorded in a specialised diary. Diary evaluations and learning modules on dysmenorrhoea and other relevant topics promote understanding of the condition and self-efficacy. An intelligent evaluation suggests suitable evidence-based and appropriate exercises. In the learning modules, patients can learn about the menstrual cycle, menstrual pain and self-management methods in a structured way. For example, there are structured courses on physiotherapy, yoga, stress reduction and relaxation methods such as progressive muscle relaxation and autogenic training.
  Arms: Intervention group

SUMMARY:
The pilot study investigates the influence of a dysmenorrhoea app on the quality of life and symptoms of women with dysmenorrhoea. The intervention group can use the app over the study period of 12 weeks in addition to usual care, while the control group only receives the usual standard care. The aim is to evaluate the effectiveness of the app and to gain insights for the design of future studies. The study is expected to last seven months and include 100-200 participants.

DETAILED DESCRIPTION:
The pilot study aims to investigate the effect of a dysmenorrhoea app on the quality of life and symptoms of women with dysmenorrhoea. Dysmenorrhoea, defined as painful menstruation, is a widespread and distressing health problem that can significantly affect the quality of life and well-being of affected women. Research into digital health applications has shown the potential to provide innovative solutions to improve care and self-management of chronic conditions.

The present study is designed as a single-blind, two-arm, randomised controlled trial in which participants will either receive the dysmenorrhoea app over a 12-week period in addition to usual care (intervention group) or only usual care as typically available (control group). The study will be conducted online. The aim is to evaluate the effectiveness of the app by analysing various questionnaires as endpoints, which were completed at T0 (baseline) and after 4 (T1), 8 (T2) and 12 weeks (T3).

The DSI, MDQ, VAS pain, FSS, FESS, PDI and DASS-21 questionnaires are defined as endpoints. The difference between the intervention group and the control group is compared in terms of the changes (change score) between the time points T0 (baseline) and T3 (post-treatment: twelve weeks). The aim was to show the superiority of the intervention. The evaluation was carried out additionally at the time points T0 and T1 (4 weeks after the start of the study) and T0 and T2 (8 weeks after the start of the study).

The hypotheses for the individual endpoints are defined as follows, whereby the respective hypothesis is to be analysed using an ANCOVA with baseline values as covariates:

Null hypothesis (H0): There is no difference between the intervention group and the control group.

Alternative hypothesis (HA): There is a difference between the intervention and control group.

In addition, this study should provide important insights for the planning of future studies. This includes aspects such as the selection of suitable endpoints, hypothesis formation and statistical analysis methods.

The planned duration of the study is expected to be seven months, starting in February 2024 and ending in August 2024. The study intends to enrol between 100 and 200 participants, aiming for an adequate sample size to ensure statistically significant results.

Overall, this pilot study is expected to provide important insights into whether and to what extent a dysmenorrhoea app can have a positive impact on the quality of life and symptoms of women with dysmenorrhoea. These results may not only help to improve patient care, but also lay the foundation for further research activities in the field of digital health applications and gynaecological health.

ELIGIBILITY:
Inclusion Criteria:

* Legal capacity
* Resident in Germany
* Female
* Age ≥18 years of age
* Known and medically confirmed dysmenorrhoea
* Ownership of an internet-enabled mobile phone and ability to use it
* Internet access for the app application and questionnaire
* Answering email address for registration
* Willingness to complete questionnaires online
* Motivation to use the app regularly
* Sufficient knowledge of the German language
* Absence of exclusion criteria

Exclusion Criteria:

* Pregnancy existing at the time of interview
* Gynaecological abdominal surgery planned in the next 12 weeks or gynaecological abdominal surgery performed within the last 8 weeks before study start
* Previous or existing access to the Endo app or other comparable digital health applications or current active prescription
* Current participation in other clinical studies
* Non-compliance with inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Dysmenorrhea Symptom Interference Scale (DSI) | 12 weeks
  Questionnaire
Moos Menstrual Distress Questionnaire, Form C (MDQ) | 12 weeks
  Questionnaire
Visual analog scale (VAS) | 12 weeks
  Questionnaire
Depression Anxiety Stress Scale mit 21 Items (DASS-21) | 12 weeks
  Questionnaire
German Version of Pain Self-Efficacy Questionnaire (FESS) | 12 weeks
  Questionnaire
Fatigue Severity Scale (FSS) | 12 weeks
  Questionnaire
Pain Disability Index (PDI) | 12 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rohloff, Dr. med., Principal Investigator — Endo Health GmbH

IPD SHARING:
Plan to Share IPD: No
There will be no sharing of individual participant data to other researchers.